CLINICAL TRIAL: NCT01621984
Title: The Evaluation of Therapeutic Riding in Children and Adolescent With Kinetic Deficits Because of Neuromuscular Disease.
Brief Title: Therapeutic Riding and Neuromuscular Disease
Acronym: TR NMD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Ioannina (Other)
Responsible Party: Principal Investigator, Avraam Ploumis, Assistant Professor of PMR, Orthopaedic Spine Surgeon, University of Ioannina
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 274/21-9-2011
Record Dates: First submitted 2012-06-12; First posted 2012-06-18 (Estimated); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: Neuromuscular Disease
Keywords: Cerebral palsy; brain injury; spinal cord injuries; muscular disease
MeSH Terms: conditions — Neuromuscular Diseases; Cerebral Palsy; Brain Injuries; Spinal Cord Injuries; Muscular Diseases | interventions — Equine-Assisted Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Therapeutic Riding/ Hippotherapy (Experimental): 12 week Therapeutic Riding program that focused on gross motor function, gross motor performance, balance, spasticity, posture and quality of life
  Interventions: Other: Therapeutic Riding/ Hippotherapy Intervention
- without Therapeutic Riding/ Hippotherapy (No Intervention)

INTERVENTIONS:
Other: Therapeutic Riding/ Hippotherapy Intervention — The Therapeutic Riding exercise intervention consisted exercises for warm up,transitions on the horseback, stretching exercises and exercises to strengthen muscles of trunk and four limps, games with balls and rings and walking of the horse to change directions as diagonal / lateral changes, cycles with open and closed eyes.
  Other Names: therapeutic riding/hippotherapy
  Arms: Therapeutic Riding/ Hippotherapy

SUMMARY:
The purpose of this current prospective study is to assess the effects of a Therapeutic Riding exercise program conducted in patients suffering from neuromuscular disease. The exercise intervention aims at improving gross motor function, gross motor performance, balance, spasticity, posture and quality of life. Patients were randomized according to age, sex, mental ability and gross motor function. Furthermore, patients will be subdivided into categories of central nervous system (brain/ spinal cord) and peripheral (peripheral nerve or muscle) diseases. The exercise program duration will be 12 weeks, once a week with 30-40 minutes sessions. Six measurements will be conducted: the Gross Motor Function Measure, the Gross Motor Performance Measure, the Quality of life Questionnaire for Children, the Pediatric Balance Scale, the dynamic plate in combination with x-ray for posture control, the Modified Ashworth Scale for spasticity and the Wisc 3 for mental ability. The results will be collected and evaluated using the statistical programme SPSS.

ELIGIBILITY:
Inclusion Criteria:

* Children with neuromuscular disease
* Parental consent
* Sitting posture capability
* Hip abduction capability on horseback
* Ability to communicate and collaborate with the researcher

Exclusion Criteria:

* Children with Scheuermann disease
* uncontrolled seizures (A) child with generalized seizure over 2 minutes in the last three months (B) Children who are not well-adjusted levels of antiepileptic drugs.
* musculoskeletal disorder that may be aggravated by the movement of the horse such as atlantoaxial instability, osteoporosis etc.
* Scoliosis > 30 degree
* Allergy to dust

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in posture control at different time points | Measures will be done: 1 two months before treatment, 2 one month before treatment, 3 one day before start of treatment, 4 six weeks after the start of treatment, 5 twelve weeks, the end of treatment 6 two months after the end of treatment.
  posture control measured by the dynamic plate in combination with x-ray.
Change from baseline in balance at different time points | Measures will be done: 1 two months before treatment, 2 one month before treatment, 3 one day before start of treatment, 4 six weeks after the start of treatment, 5 twelve weeks, the end of treatment 6 two months after the end of treatment.
  Balance measured by the Pediatric Balance Scale

SECONDARY OUTCOMES:
Improvement in Gross Motor Function | Measures will be done: 1 two months before treatment, 2 one month before treatment, 3 just before treatment, 4 six weeks after the start of treatment, 5 twelve weeks, the end of treatment 6 two months after the end of treatment.
  Gross Motor Function measured by the Gross Motor Function Measure (GMFM)
Improvement in Gross Motor Performance | Measures will be done: 1 two months before treatment, 2 one month before treatment, 3 just before treatment, 4 six weeks after the start of treatment, 5 twelve weeks, the end of treatment 6 two months after the end of treatment.
  Gross Motor Performance measured by the Gross Motor Performance Measure (GMPM)
Decrease of spasticity | Measures will be done: 1 two months before treatment, 2 one month before treatment, 3 just before treatment, 4 six weeks after the start of treatment, 5 twelve weeks, the end of treatment 6 two months after the end of treatment.
  Spastisity measured by the Modified Ashworth Scale
Improvement in Quality of life | Measures will be done: 1 two months before treatment, 2 one month before treatment, 3 just before treatment, 4 six weeks after the start of treatment, 5 twelve weeks, the end of treatment 6 two months after the end of treatment.
  Quality of life measured by the Quality of life Questionnaire for Children

CONTACTS AND LOCATIONS:
Overall Officials: Avraam Ploumis, Principal Investigator — University Hospital, Ioannina
Locations (1):
- University Hospital of Ioannina, Ioannina, Greece